CLINICAL TRIAL: NCT04763421
Title: A Prospective, Single-Arm Multi-Center Study of the ENSEAL X1 Curved Jaw Tissue Sealer and Generator G11 in Upper Gastrointestinal, Lower Gastrointestinal, and Gynecological Procedures
Brief Title: A Prospective, Single-Arm Multi-Center Study of the ENSEAL X1 Curved Jaw Tissue Sealer in Select Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG_2019_01
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Upper GI; Lower GI; Gynecological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Upper Gastrointestinal/Lower Gastrointestinal/Gynecological (Experimental): Any upper gastrointestinal/lower gastrointestinal/gynecological procedure where the ENSEAL X1 Curved Jaw is used for vessel transection according to instructions for use.
  Interventions: Device: ENSEAL X1 Curved Jaw

INTERVENTIONS:
Device: ENSEAL X1 Curved Jaw — ENSEAL X1 Curved Jaw is used for vessel transection according to instructions for use.

SUMMARY:
This prospective, single-arm, multi-center study will collect clinical data in a post-market setting by procedure group (upper gastrointestinal [GI], lower GI, and gynecological). Investigators will perform each procedure using the device in compliance with their standard surgical approach and the ENSEAL X1 Curved Jaw and Generator G11 instructions for use.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the acceptable performance and safety of the ENSEAL X1 Curved Jaw and Generator G11 devices when used per the instructions for use.

ELIGIBILITY:
Inclusion Criteria:

1. Primary laparoscopic or open procedure (upper gastrointestinal, lower gastrointestinal, or gynecological) where at least one vessel is planned to be transected by the ENSEAL X1 Curved Jaw device per the instructions for use;
2. Willingness to give consent and comply with all study-related evaluations and visit schedule; and
3. At least 18 years of age.

Exclusion Criteria:

1. Physical or psychological condition which would impair study participation; or
2. Enrollment in a concurrent interventional clinical study that could impact the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmar Shah, MD, Principal Investigator — Yeovil District Hospital; Anna Fagotti, MD, Principal Investigator — Gemelli Hospital; Sergio Alfieri, MD, Principal Investigator — Gemelli Hospital; Richard Skipworth, MD, Principal Investigator — Royal Infirmary of Edinburgh; Hugh Paterson, MD, Principal Investigator — Western General Hospital; Keith Gersin, MD, Principal Investigator — Wake Forest University Health Sciences; James Hopkins, MD, Principal Investigator — Southmead Hospital
Locations (6):
- Atrium Health, Charlotte, North Carolina, United States
- Gemelli Hospital, Rome, Italy
- United Kingdom (4):
  - Southmead Hospital, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- ENSEAL X1 Curved Jaw: All participants were treated with ENSEAL X1 curved jaw device for transection of at least one vessel during laparoscopic or open procedure (upper gastrointestinal [GI], lower GI, or gynecological).
Period: Overall Study
Arm/Group | ENSEAL X1 Curved Jaw
Started | 145
Completed | 145
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.28 (15.904)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 135
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 133
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Vessels With Less Than or Equal to (<=) Grade 3 Hemostasis Based on Hemostasis Grading Scale
Description: Number of vessels with <= Grade 3 hemostasis based on hemostasis grading scale were reported. A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with ENSEAL X1; or Grade 4: significant bleeding (example, pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (example, hemoclips, staples, sutures, fibrin sealants, other advanced energy products).
Time Frame: On the day of transection (Day 0)
Population: Full Analysis Set (FAS) included participants for whom the ENSEAL X1 device was utilized during the surgical procedure. Here, the number of vessels transected analyzed included all vessels that were transected and analyzed for this outcome measure.
Measure: Count of Units; unit: Vessels transected
Units Other Than Participants: Vessels transected
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 145
Number analyzed (Vessels transected) | 279
Vessels transected | 279

2. Primary Outcome: Number of Participants With Device-related Adverse Events (AEs)
Description: Number of participants with device-related AEs were reported. Device-related AEs were those AEs identified as having a relationship of possibly, probably, or causally with the study devices.
Time Frame: From Day 0 up to post-procedure follow up visit (up to 28 days)
Population: The Safety Analysis Set (SAS) included all participants who signed informed consent and for whom the ENSEAL X1 device was utilized during the surgical procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 145
Participants | 2

3. Secondary Outcome: Number of Participants With Adhesion Removal or Division Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Number of participants with adhesion removal or division using ENSEAL X1 device as assessed by Surgeon Satisfaction scale score were reported. Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for adhesion removal or division by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: FAS included participants for whom the ENSEAL X1 device was utilized during the surgical procedure. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 49
Participants
  Very Dissatisfied | 0
  Dissatisfied | 0
  Neither Satisfied or Dissatisfied | 1
  Satisfied | 27
  Very Satisfied | 21

4. Secondary Outcome: Number of Participants With Lymphatics Bundles Division Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Number of participants with lymphatics bundles division using ENSEAL X1 device as assessed by Surgeon Satisfaction scale score were reported. Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for lymphatic bundles by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 27
Participants
  Very Dissatisfied | 0
  Dissatisfied | 0
  Neither Satisfied or Dissatisfied | 1
  Satisfied | 18
  Very Satisfied | 8

5. Secondary Outcome: Number of Participants With Tissues Bundles Division Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Number of participants with tissues bundles division using ENSEAL X1 device as assessed by Surgeon Satisfaction scale score were reported. Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissues bundles by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 55
Participants
  Very Dissatisfied | 0
  Dissatisfied | 0
  Neither Satisfied or Dissatisfied | 1
  Satisfied | 26
  Very Satisfied | 28

6. Secondary Outcome: Number of Participants With Tissues Grasping Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Number of participants with tissues grasping using ENSEAL X1 device as assessed by Surgeon Satisfaction scale score were reported. Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissues grasping by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 67
Participants
  Very Dissatisfied | 0
  Dissatisfied | 4
  Neither Satisfied or Dissatisfied | 9
  Satisfied | 31
  Very Satisfied | 23

7. Secondary Outcome: Number of Participants With Tissues Cutting Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Number of participants with tissues cutting using ENSEAL X1 device as assessed by Surgeon Satisfaction scale score were reported. Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissues cutting by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 87
Participants
  Very Dissatisfied | 1
  Dissatisfied | 1
  Neither Satisfied or Dissatisfied | 3
  Satisfied | 38
  Very Satisfied | 44

8. Secondary Outcome: Number of Participants With Tissues Dissection Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Number of participants with tissues dissection using ENSEAL X1 device as assessed by Surgeon Satisfaction scale score were reported. Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissues dissection by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 107
Participants
  Very Dissatisfied | 0
  Dissatisfied | 0
  Neither Satisfied or Dissatisfied | 3
  Satisfied | 59
  Very Satisfied | 45

9. Secondary Outcome: Number of Vessels With Hemostasis (Grade 1 to 4) Based on Hemostasis Grading Scale
Description: Number of vessels with hemostasis (Grade 1 to 4) based on hemostasis grading scale were reported. A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with ENSEAL X1; or Grade 4: significant bleeding (example, pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (example, hemoclips, staples, sutures, fibrin sealants, other advanced energy products).
Time Frame: On the day of transection (Day 0)
Population: FAS included participants for whom the ENSEAL X1 device was utilized during the surgical procedure. Here, the number of vessels transected analyzed included all vessels that were transected and analyzed for this outcome measure.
Measure: Count of Units; unit: vessels transected
Units Other Than Participants: vessels transected
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 145
Number analyzed (vessels transected) | 279
vessels transected
  Grade 1 | 258
  Grade 2 | 12
  Grade 3 | 9
  Grade 4 | 0

10. Secondary Outcome: Percentage of Grade 4 Vessel Transections Requiring Hemostasis Measures
Description: Percentage of Grade 4 vessel transections requiring hemostasis measures were planned to be reported. Data was not collected and analyzed for this outcome measure because there were no hemostatic grade 4 vessel transections.
Time Frame: On the day of transection (Day 0)
Population: FAS included participants for whom the ENSEAL X1 device was utilized during the surgical procedure.
Units Other Than Participants: percentage of vessels transected
Arm/Group | ENSEAL X1 Curved Jaw
Number analyzed (Participants) | 0
Number analyzed (percentage of vessels transected) | 0

ADVERSE EVENTS:
Time Frame: From Day 0 up to post-procedure follow up visit (Up to 28 days)
Description: The Safety Analysis Set (SAS) included all participants who signed informed consent and for whom the ENSEAL X1 device was utilized during the surgical procedure.
Arm/Group | ENSEAL X1 Curved Jaw
All-Cause Mortality (participants affected / at risk) | 0/145
Serious Adverse Events (participants affected / at risk) | 10/145
Other Adverse Events (participants affected / at risk) | 58/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENSEAL X1 Curved Jaw (N=145)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphatic fistula (Vascular disorders) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENSEAL X1 Curved Jaw (N=145)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 21 (21)
Vomiting (Gastrointestinal disorders) | 10 (10)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Pain (General disorders) | 14 (14)
Pyrexia (General disorders) | 4 (4)
Cystitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Genital contusion (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 3 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 10 (10)
Wound complication (Injury, poisoning and procedural complications) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Hallucination (Psychiatric disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04763421/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT04763421/SAP_001.pdf